CLINICAL TRIAL: NCT03758066
Title: PlusCare: Mobile Platform to Increase Linkage to Care in Adolescents Living With HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dimagi Inc. (Industry)
Collaborators: Boston Children's Hospital (Other); Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 9R44MH117956-02 (NIH)
Record Dates: First submitted 2018-11-09; First posted 2018-11-29 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: HIV/AIDS
Keywords: youth; young adults; digital health; mobile application; case management
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Pre-post quasi-experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PlusCare (Other): Patients and case managers who work with them will be given access to a web-/mobile-based application, PlusCare, to support various case management activities for one year.
  Interventions: Device: PlusCare

INTERVENTIONS:
Device: PlusCare — PlusCare is a mobile application designed to be used by youth and young adults with HIV and case managers.

SUMMARY:
While major advancements in medical technology over the past decade have significantly improved the life expectancy of persons infected with human immunodeficiency virus (HIV), HIV-positive youth today face new barriers to the treatment of HIV as a chronic, manageable illness. The mobile system proposed will help improve linkage to care through mobile technology support for the case management of youth living with HIV. Results of this project will determine the impact of this system on case management processes and outcomes and have implications for the care of youth living with other chronic, complex illnesses.

DETAILED DESCRIPTION:
With the advancement of medical treatments, which has contributed to the overall decrease in opportunistic infections and deaths related to human immunodeficiency virus (HIV) in youth, there is a need to ensure that youth living with HIV (YLH) are linked to and engaged in care to successfully achieve viral suppression. While an increasing number of mobile health (mHealth) technologies have been designed to address HIV prevention and care, a critical gap in innovation remains in tools designed to address the specific needs of YLH. In a Phase I project, investigators demonstrated the acceptability and feasibility of a user-centered prototype design of PlusCare, an mHealth application that can be used by YLH and their case managers (CMs) to support HIV care. Results of Phase I suggest that PlusCare could facilitate multi-disciplinary, team-based case management of YLH by supporting the sharing and signing of documents remotely, automation of adherence reminders, sharing of lab results, alerts CMs about program requirements related to age and developmental milestones, streamlining of communication between multiple members of a patient's case management team and the patient, and offering accessibility to data from multiple modalities. In this Phase II project, investigators will conduct a mixed methods, non-randomized pre-post study with CMs (N=20) and YLH patients (N=70) to examine the use of PlusCare on case management processes and health outcomes (i.e., HIV viral load, medical visit frequency and gaps) in 3 different case management programs at 2 different clinical study site settings. An initial cost analysis will be performed to assess potential cost effectiveness. Results of these Phase I and II projects will inform the development of a product that can be used in multiple case management settings and prepare PlusCare for future commercialization. Results have implications for future development of PlusCare to serve the broader HIV population (YLH aged 25-34 years old and at-risk individuals) as well as youth living with other chronic health conditions.

ELIGIBILITY:
PATIENTS:

Inclusion Criteria:

* between 13-25 years old
* HIV positive
* enrolled in treatment at a participating study site
* owns or has ability to access a smartphone (e.g., iPhone, Android) for one year

Exclusion Criteria:

* Non-English speaker or
* Visually/hearing impaired

CASE MANAGERS:

Inclusion Criteria:

* Actively employed at a participating study site
* Performs case management duties with HIV-positive patients aged 13-25 years.

Exclusion Criteria:

* (None)

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan L Jackson, MEng, Principal Investigator — Dimagi Inc.; Vikram S Kumar, MD, Principal Investigator — Dimagi Inc.
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guss, CE, Woods, ER, Cooper, ER, Burchett, S, Fuller, JM, Dumont, O, Ho, YX, Robinson, M, Swendeman, D, Haberer, J, Mulvaney, S, & Kumar, V. (2020). PlusCare: A Mobile Platform Designed to Increase Linkage to Care for Youth Living with HIV/AIDS. J Adol Health, 66(2),127-128. doi:https://doi.org/10.1016/j.jadohealth.2019.11.255 (Abstract)
- [Result] Fee C, Fuller J, Guss CE, Woods ER, Cooper ER, Bhaumik U, Graham D, Burchett SK, Dumont O, Martey EB, Narvaez M, Haberer JE, Swendeman D, Mulvaney SA, Kumar VS, Jackson JL, Ho YX. A Digital Platform to Support HIV Case Management for Youth and Young Adults: Mixed Methods Feasibility Study. JMIR Form Res. 2022 Nov 21;6(11):e39357. doi: 10.2196/39357. PMID 36409541

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited and enrolled into the study between January 2019 to June 2019 from 3 HIV/AIDS programs at two large, private, not-for-profit academic hospitals in the metro Boston area. Participants were case management program team members (CMs) and adolescents and young adults (AYA) living with HIV. CMs were enrolled and trained on the system first. Patients were then enrolled on a rolling basis. An RA at each site assessed eligibility, consented and enrolled participants.
Pre-assignment Details: There were no significant effects that occurred after participant enrollment that affected enrolled participants receiving the intervention. This was a one-armed prospective study where participants were enrolled into the study and then enrolled into the PlusCare system in-person in one session.
Groups:
- PlusCare: AYA living with HIV and CMs who work with them will be given access to a web-/mobile-based application, PlusCare, to support various case management activities for one year. PlusCare is a web/mobile application designed to be used by youth and young adults with HIV and case managers.
Period: Overall Study
Arm/Group | PlusCare
Started | 65 (20 CMs and 45 AYA living with HIV were enrolled)
Completed | 51 (13 CMs and 38 AYA living with HIV completed all study activities)
Not Completed | 14
Not completed — Lost to Follow-up | 14

BASELINE CHARACTERISTICS:
Population: Participants were members of HIV case management care team members (CMs) in 3 different programs and adolescent and young adult (AYA) patients living with HIV who they work with in the programs.
Arm/Group | PlusCare
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants] — Population: Demographics are reported for each of the 2 participant types (CM and AYA living with HIV)
  Participants
    AYA living with HIV: number analyzed (Participants) | 45
    AYA living with HIV: <=18 years | 12
    AYA living with HIV: Between 18 and 65 years | 33
    AYA living with HIV: >=65 years | 0
    CM: number analyzed (Participants) | 20
    CM: <=18 years | 0
    CM: Between 18 and 65 years | 20
    CM: >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographics are reported for each of the 2 participant types (CM and AYA living with HIV)
  Participants
    AYA living with HIV: number analyzed (Participants) | 45
    AYA living with HIV: Female | 23
    AYA living with HIV: Male | 22
    CM: number analyzed (Participants) | 20
    CM: Female | 18
    CM: Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Demographics are reported for each of the 2 participant types (CM and AYA living with HIV)
  Participants
    AYA living with HIV: number analyzed (Participants) | 45
    AYA living with HIV: Hispanic/Latino | 8
    AYA living with HIV: Not Hispanic, White | 4
    AYA living with HIV: Not Hispanic, Black | 24
    AYA living with HIV: Not Hispanic, Other (incl. Native American, Asian/Pacific Islander, More than one) | 6
    AYA living with HIV: Unknown ethnicity | 3
    CM: number analyzed (Participants) | 20
    CM: Hispanic/Latino | 1
    CM: Not Hispanic, White | 12
    CM: Not Hispanic, Black | 4
    CM: Not Hispanic, Other (incl. Native American, Asian/Pacific Islander, More than one) | 1
    CM: Unknown ethnicity | 2
Education [Count of Participants; unit: Participants] — Population: Demographics are reported for each of the 2 participant types (CM and AYA living with HIV)
  Participants
    AYA living with HIV: number analyzed (Participants) | 44
    AYA living with HIV: High school graduate or less | 24
    AYA living with HIV: Some college credit or more | 20
    AYA living with HIV: Bachelor's Degree | 0
    AYA living with HIV: Master's Degree | 0
    AYA living with HIV: Doctoral Degree | 0
    AYA living with HIV: Professional Degree | 0
    CM: number analyzed (Participants) | 20
    CM: High school graduate or less | 0
    CM: Some college credit or more | 0
    CM: Bachelor's Degree | 7
    CM: Master's Degree | 7
    CM: Doctoral Degree | 4
    CM: Professional Degree | 2
Smartphone ownership [Count of Participants; unit: Participants] — Population: Demographics are reported for each of the 2 participant types (CM and AYA living with HIV)
  Participants
    AYA living with HIV: number analyzed (Participants) | 45
    AYA living with HIV: iPhone | 40
    AYA living with HIV: Android | 5
    CM: number analyzed (Participants) | 20
    CM: iPhone | 17
    CM: Android | 3
Hours on the phone per day [Count of Participants; unit: Participants] — Population: Demographics are reported for each of the 2 participant types (CM and AYA living with HIV)
  Participants
    AYA living with HIV: number analyzed (Participants) | 45
    AYA living with HIV: 0-3 hours | 8
    AYA living with HIV: 4-6 hours | 19
    AYA living with HIV: 7+ hours | 18
    CM: number analyzed (Participants) | 20
    CM: 0-3 hours | 9
    CM: 4-6 hours | 8
    CM: 7+ hours | 3
Tech savvy [Mean (Standard Deviation); unit: units on a scale] — Survey item: How tech savvy would you rate yourself, from 1 to 10? (1=not savvy, 10=very savvy) Population: Demographics are reported for each of the 2 participant types (CM and AYA living with HIV)
  units on a scale
    AYA living with HIV: number analyzed (Participants) | 45
    AYA living with HIV | 7.86 (1.58)
    CM: number analyzed (Participants) | 20
    CM | 7.05 (1.23)

OUTCOME MEASURES:

1. Primary Outcome: CD4 Cell Count
Description: Comparison of average CD4 cell count (cells/mm^3) between pre and post time points
Time Frame: 1 year prior to baseline (pre), 1 year post-baseline (post)
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Groups:
- PlusCare: AYA living with HIC given access to a web-/mobile-based application, PlusCare, to support various case management activities for one year
Arm/Group | PlusCare
Number analyzed (Participants) | 45
cells/mm^3
  Pre | 996 [857 to 1157]
  Post | 1049 [898 to 1224]

2. Primary Outcome: Viral Load
Description: Comparison of average viral load (copies/mL) between pre and post time points
Time Frame: 1 year prior to baseline (pre), 1 year post-baseline (post)
Measure: Mean (95% Confidence Interval); unit: copies/mL
Groups:
- PlusCare: AYA living with HIV given access to a web-/mobile-based application, PlusCare, to support various case management activities for one year.
Arm/Group | PlusCare
Number analyzed (Participants) | 45
copies/mL
  Pre | 32.0 [17.9 to 60.4]
  Post | 24.7 [12.1 to 47.9]

3. Primary Outcome: Appointment Adherence Rate
Description: Comparison of median appointment adherence ratio between pre and post time points, i.e., (Actual completed appointments) / (Expected appointments) where expected appointments includes completed appointments, no shows, and cancellations
Time Frame: 1 year prior to baseline (pre), 1 year post-baseline (post)
Measure: Median (Standard Deviation); unit: appointment adherence ratio
Groups:
- PlusCare: AYA living with HIV participants given access to a web-/mobile-based application, PlusCare, to support various case management activities for one year.
Arm/Group | PlusCare
Number analyzed (Participants) | 45
appointment adherence ratio
  Pre | 0.60 (.19)
  Post | .67 (.25)

4. Secondary Outcome: Proximal Outcomes (Monthly Medication Adherence Item)
Description: Self-reported levels of medication adherence were reported on a monthly basis, where AYA living with HIV rated their adherence to their prescribed medication using the self-rating scale item (SRSI) single-item adherence measure. Patients reported medication adherence for the past month on a 6-point Likert scale ranging from 1 ("very poor") to 6 ("excellent"). Patients received monthly SMS text messages alerting them to report adherence via survey forms created in the PlusCare app. Mean self-reported monthly medication adherence ratings across 12 months is reported.
Time Frame: Monthly
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PlusCare
Number analyzed (Participants) | 45
score on a scale | 4.7 (.23)

5. Secondary Outcome: Patient-centered Outcomes (Quality of Life): Self-reported Responses to Survey
Description: Self-reported scores to the General Health item of the CDC "Health Days Measure" Core Module (CDC HRQOL-4) item were compared between 3 timepoints, with scores ranging from 1 ("Poor") to 5 ("Excellent").
Time Frame: 1 year (Baseline, 6-month, 12-month)
Population: Participants who completed the quality of life general health assessment (CDC HRQOL-4) at baseline, 6 months, and 12 months (end of study).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PlusCare
Number analyzed (Participants) | 45
score on a scale
  Baseline | 3.6 (.12)
  6-month | 3.6 (.16)
  12-month | 3.9 (.16)
Statistical Analysis 1: Comparison: PlusCare; A two-tailed non-parametric one-sample paired sign test was used to determine whether to reject or fail to reject the null hypothesis that the mean difference of scores between any of the 2 of 3 timepoints is 0 (Baseline v. 6-month, 6-month v. 12-month, and Baseline v. 12-month); Test type: Other; p = .03, Sign test — P-value reported for quality of life measured between baseline and 12-month follow-up with a statistical significance threshold of .05

6. Secondary Outcome: Patient-centered Outcomes (Self-efficacy): Self-reported Responses to Survey
Description: Self-reported average scores to the Self-Efficacy for Managing Chronic Disease 6-item Scale (SEMCD6) were compared between 3 timepoints. SEMCD6 scores range from 1 to 10, with higher numbers indicating higher self-efficacy.
Time Frame: 1 year (Baseline, 6-month, 12-month)
Population: Participants who completed self-efficacy assessment (SEMCD6) at baseline, 6 months, and 12 months (end of study).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PlusCare
Number analyzed (Participants) | 45
score on a scale
  Baseline | 7.8 (.3)
  6-month | 7.8 (.36)
  12-month | 8.6 (.27)
Statistical Analysis 1: Comparison: PlusCare; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = .02, Sign test — P-value reported for self-reported self-efficacy in chronic disease management between baseline and 12-month follow-up with a statistical significance threshold of .05
Statistical Analysis 2: Comparison: PlusCare; Test type: Other; p = .02, Sign test — P-value reported for self-reported self-efficacy in chronic disease management between 6- and 12-month follow-up with a statistical significance threshold of .05

7. Secondary Outcome: System Usability (User Satisfaction): System Usability Scale
Description: Self-reported ratings of perceived system usability on the 10-point Likert-scaled System Usability Scale (SUS) scored in a range of 0 of 100, with higher scores indicating higher usability, were collected at end of study.
Time Frame: 1 year
Population: Summary of SUS scores reported for 13 (out of 20) CMs and 38 (out of 45) AYA living with HIV participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PlusCare
Number analyzed (Participants) | 51
score on a scale
  AYA living with HIV: number analyzed (Participants) | 38
  AYA living with HIV | 63 (10.6)
  CM: number analyzed (Participants) | 13
  CM | 51 (7.9)

ADVERSE EVENTS:
Time Frame: Approximately 1 year from enrollment
Description: Adverse events (AE) in this study will be any breach of confidentiality. A serious AE will be considered to have occurred if a subject's identity or personal health information becomes known to someone who is not supposed to have (and previously did not have) access to the information.
Arm/Group | PlusCare
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03758066/Prot_SAP_000.pdf